CLINICAL TRIAL: NCT05914311
Title: Use of Dermabond in Mitigation of Spinal Cord Stimulation Trial Lead Migration
Brief Title: Use of Dermabond in Mitigation of Spinal Cord Stimulation (SCS) Trial Lead Migration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00087042
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain
Keywords: Spinal Cord Stimulation (SCS); chronic pain; stimulator
MeSH Terms: conditions — Chronic Pain | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Suture Group (Active Comparator): secure one of the 2 trial leads with suture only-randomized to left or right
  Interventions: Device: Suture
- Dermabond (Experimental): secure one of the 2 trial leads to be secured with both dermabond and suture-randomized to left or right
  Interventions: Device: Suture; Device: Dermabond

INTERVENTIONS:
Device: Suture — secures SCS trial leads with a suture
Device: Dermabond — secures SCS trial leads with dermabond
  Arms: Dermabond

SUMMARY:
During the typical SCS trial the leads remain outside of the skin and can be prone to migration. The leads are typically secured in place with suture, tape, or a combination of both. This study will evaluate the amount of movement based on the method of being secured at the time of placement

DETAILED DESCRIPTION:
Spinal Cord stimulator trials require precise placement of leads to get appropriate distribution of pain.1 Since the leads are not anchored into the tissue, migration of the leads can occur and result in suboptimal trial. Migration (or movement in the epidural space after placement) of the leads can result in up to 2.49 mm to 3.24 mm migration in the leads depending on trial length . During the trial the leads remain outside of the skin and can be prone to migration. The leads are typically secured in place with suture, tape, or a combination of both. This study will evaluate the amount of movement based on the method of being secured at the time of placement

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18
* having a spinal cord stimulator trial lead placement done
* lead placement to be done in the thoracic spine area

Exclusion Criteria:

* dermabond allergy
* inability to place 2 leads in subject
* lead placement not in thoracic spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Migration rate of trial leads | From Baseline through Day 8
  Migration rate of trial leads anchored with Dermabond and suture versus suture alone will be measured by change in trial lead position as measured in millimeters when comparing initial x-ray after placement versus x-ray taken at lead removal 5-8 days after placement

SECONDARY OUTCOMES:
Patient Satisfaction Score | Day 8
  Patient satisfaction score will be valued on a 0-10 scale, with 0-not satisfied at all up to 10-greatest level of satisfaction
Rate of Infection | Day 8
  determine if a longer trial predisposes spinal cord stimulation trial lead insertion site to a higher rate of infection
Difference in Lead Position - Prone Fluoroscopy vs Upright X-ray | Day 8
  Difference in lead position on prone (face down) fluoroscopy vs upright (standing) x-ray
Number of Patients with Pain Relief | Day 8
  Number of patients who received pain relief from the spinal cord stimulation trial. Number of responders to the prognostic lead placements defined as >50% pain relief over the length of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Carlyle Hamsher, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
analysis will include all participant data via publication

DOCUMENTS (1):
  • Informed Consent Form (2025-04-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT05914311/ICF_000.pdf